CLINICAL TRIAL: NCT04971122
Title: Comparison of the Effects of Trendelenburg Position and Passive Leg Lift on Hemodynamics in Abdominal Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yangmi
Record Dates: First submitted 2021-06-20; First posted 2021-07-21 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: The Angle of Trendelenburg

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trendeleburg -5 degree group,-10 degree group,-15 degree group (Other): Norepinephrine was continuously pumped at 0.5ug/kg/min
  Interventions: Other: Trendeleburg -5 degree,-10 degree,-15 degree

INTERVENTIONS:
Other: Trendeleburg -5 degree,-10 degree,-15 degree — Use a -5 or -10 or -15 degree trendelenburg position

SUMMARY:
How to maintain the stability of circulation during anesthesia has always been a concern of clinicians, including shorting the preoperative fasting time under the condition of full preoperative preparation, and giving appropriate amount of nutrient solution in combination with the patient's situation 2~4 h before surgery to reduce the blood volume insufficiency of patients before general anesthesia induction, vasoactive drugs, etc. Among them, passive leg lifting experiment is widely recognized in the world. Although passive leg lifting has many advantages, it still has some limitations in the operation process. This study tried to find the corresponding head low and foot high Angle corresponding to the same hemodynamic changes caused by passive leg lifting.

DETAILED DESCRIPTION:
For low head and high feet, studies have shown that 20° can reduce the incidence of hypotension during the induction period of general anesthesia in patients undergoing gastrectomy and has therapeutic effect on it, as well as reduce the use of vasoactive drugs during the induction period of general anesthesia. There were no perioperative complications.

The passive leg lift test can be repeated and does not overload the patient with fluid. However, there is no relevant research on the relationship between the two, which is exactly the innovation of this topic.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75 years old
* Good image of TTE can be obtained
* Sedative mechanical ventilation （Vt 8～10ml/kg）
* Circulation was relatively stable before the experiment began
* There is no contraindication to rehydration

Exclusion Criteria:

* TTE acquisition is not ideal
* Patients did not agree to participate in the experiment
* Diseases of the central nervous system，patients with increased intracranial pressure
* Arrhythmia patients;
* Patients with increased intra-abdominal pressure;
* Bedridden patients;
* Patients with venous thrombosis of lower limbs;
* Patients with venous foreign body of lower limbs;
* Patients with circulatory instability;
* Patients with obstructive shock;
* Patients with moderate or above heart valve reflux

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
PPV(pulse pressure variation) | T1:A supine position with a 10° upward bed angulation；T2: After passive leg lift；T3：The same position with T1；T4:After trendelenburg position；T5:The same position with T1;T6:After fluid infusion
  Change from PPV at T1to T6
VTI(velocity time integral) | T1:A supine position with a 10° upward bed angulation；T2: After passive leg lift；T3：The same position with T1；T4:After trendelenburg position；T5:The same position with T1;T6:After fluid infusion
  Change from VTI at T1 to T6

SECONDARY OUTCOMES:
SBP(Systolic Blood Pressure) | T1:A supine position with a 10° upward bed angulation；T2: After passive leg lift；T3：The same position with T1；T4:After trendelenburg position；T5:The same position with T1;T6:After fluid infusion
  The variation tendency of T1 to T6
MAP(Mean Artery Pressure) | T1:A supine position with a 10° upward bed angulation；T2: After passive leg lift；T3：The same position with T1；T4:After trendelenburg position；T5:The same position with T1;T6:After fluid infusion
  The variation tendency of T1 to T6
HR HR(Heart Rate) | T1:A supine position with a 10° upward bed angulation；T2: After passive leg lift；T3：The same position with T1；T4:After trendelenburg position；T5:The same position with T1;T6:After fluid infusion
  The variation tendency of T1 to T6

CONTACTS AND LOCATIONS:
Overall Officials: Dan Hua, Master, Principal Investigator — Dalian Medical University
Locations (1):
- The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No